CLINICAL TRIAL: NCT01294761
Title: Switching From Lopinavir/Ritonavir Plus Tenofovir and Emtricitabine (or Lamivudine) to Darunavir (Prezista) and Raltegravir to Evaluate Renal Function
Brief Title: Comparing Continuing Tenofovir, Emtricitabine (or Lamivudine) Plus Lopinavir and Switching to Raltegravir Plus Darunavir
Acronym: SPARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Global Health and Medicine, Japan (Other Government)
Collaborators: Ministry of Health, Labour and Welfare, Japan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FWA00005823-SPARE2011; UMIN000005116 (Other: University Hospital Medical Information Network (UMIN))
Record Dates: First submitted 2011-02-10; First posted 2011-02-11 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: HIV Infections
Keywords: HIV-1; AIDS; Clinical Trials, Randomized
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Raltegravir, Darunavir/r (Experimental): An arm to change the regimen from: Kaletra 4 tabs QD and Truvada 1 tab QD or Kaletra 4 tabs QD, Viread 1 tab QD, Epivir300mg 1 tab (or Epivir 150mg 2 tabs) QD
  to: Prezista naive 2 tabs PC QD, Norvir soft-capsule 1 cap PC QD and Isentress 1 tab BID or Prezista 2 tabs PC BID and Norvir soft-capsule 1 cap PC BID, and Isentress 1 tab BID
  Interventions: Drug: Raltegravir, Darunavir/r
- Tenofovir, Emtricitabine, Lopinavir/r (No Intervention): An arm continuing on the same regimen before the randomization as Kaletra 4 tabs QD and Truvada 1 tab QD or Kaletra 4 tabs QD, Viread 1 tab QD, Epivir300mg 1 tab (or Epivir 150mg 2 tabs) QD

INTERVENTIONS:
Drug: Raltegravir, Darunavir/r — An arm to change the regimen to: raltegravir and darunavir/ritonavir
  Prezista naive 2 tabs PC QD, Norvir soft-capsule 1 cap PC QD and Isentress 1 tab BID or Prezista 2 tabs PC BID and Norvir soft-capsule 1 cap PC BID, and Isentress 1 tab BID
  from: Kaletra 4 tabs QD and Truvada 1 tab QD or Kaletra 4 tabs QD, Viread 1 tab QD, Epivir300mg 1 tab (or Epivir 150mg 2 tabs) QD
  Other Names: NRTI sparing regimen
  Arms: Raltegravir, Darunavir/r

SUMMARY:
The main objective of this clinical trial in randomizing HIV infected patients under good HIV control with tenofovir (TDF), emtricitabine (or lamivudine) plus lopinavir/ritonavir (LPV/r) into switching the regimen to raltegravir (RAL) with darunavir/ritonavir (DRV/r) or continuing the ongoing regimen to compare these two groups' estimated glomerular filtration rate (eGFR) is to investigate whether anti-HIV treatment that does not contain TDF or other reverse-transcriptase inhibitors (NTRI sparing regimen) can be protective of patients' renal functions and has the same virological efficacy in comparison with a standard treatment with TDF, or not.

DETAILED DESCRIPTION:
Eligibility criteria are HIV infected outpatients or inpatients that are:

without history virological failure including protease inhibitors or raltegravir (disregarding whether the patient had a history of drug resistance or drug holiday, or not) taking LPV/r+TVD (or TDF+lamivudine) for longer than 15 weeks before the enrollment with HIV viral load less than 50 copies/ml for 15 weeks, including those with blips (one time episode of detectable level HIV viraemia which are proceeded and followed by undetectable viraemia).

20 years old or older Japanese willing to participate in the trial and able to agree to the informed consent. Main outcome measures are to investigate if the estimated glomerular filtration rate (eGFR) of the intervened group with RAL+DRV/r improves by 10% or more by intention to treat (ITT) analysis at the time of 48 weeks after the start of the trial.

Other outcome measures are:

virological efficacy of the group on DRV/r+RAL (after 48 weeks and up to 96 weeks) comparison of other renal function markers between the two arms: serum creatinine, urine beta-2 microglobulin, tubular resorption rate of phosphate, urine albumin, N-acetyl-beta-glucosaminidase, serum cystatin C, urine protein and urine glucose (after 48 weeks and up to 96 weeks) comparison of lipid markers between the two arms: triglycerides, HDL cholesterol, LDL cholesterol and total cholesterol (after 48 weeks and up to 96 weeks) discontinuation rate of each arm, reason and timing of the discontinuation or the treatment change up to 96 weeks adverse events of each arm, symptoms and rate up to 96 weeks blood plasma concentration level of RAL and DRV of all consented intervened cases at National Center for Global Health and Medicine

ELIGIBILITY:
Inclusion Criteria: HIV infected outpatients or inpatients that are

* without history virological failure including protease inhibitors or raltegravir (disregarding whether the patient had a history of drug resistance or drug holiday, or not)
* taking LPV/r+TVD (or TDF+lamivudine) for longer than 15 weeks before the enrollment
* with HIV viral load less than 50 copies/ml for 15 weeks, including those with blips (one time episode of detectable level HIV viraemia which are proceeded and followed by undetectable viraemia)
* 20 years old or older
* Japanese
* willing to participate in the trial and able to agree to the informed consent

Exclusion Criteria: cases applicable to any of the following will be excluded from this trial

* HBs antigen positive within 15 weeks to the enrollment (cases confirmed as HBs antibody positive can be enrolled without HBs antigen testing)
* malabsorption or gastrointestinal symptoms that affect absorption of the drugs, or dysphagia cases
* clinical data within 15 weeks before the start of the trial and of the closest date to the enrollment that are GPT 2.5 times the highest of the normal range (grade 2) or eGFR less than 60ml/min (Cockcroft-Gault formula)
* cases with opportunistic infections requiring treatment (primary and secondary preventive prophylaxis can be administrated during the study)
* cases during pregnancy or nursing period, or with a possibility for pregnancy
* using drugs that are prohibited to combine for drug interaction with the drugs of this trial
* other cases that are decided by the patient's physician as not suitable for the trial

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2011-02; Primary Completion 2012-02 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
eGFR improvement comparison of two arms by ITT analysis | 48 weeks
  To investigate whether the estimated glomerular filtration rate (eGFR) of the intervened group with RAL+DRV/r improves by 10% or more by intention to treat (ITT) analysis at the time of 48 weeks after the start of the study, or not.

SECONDARY OUTCOMES:
Virological efficacy | 48 weeks up to 96 weeks
  Virological efficacy of the group on DRV/r+RAL
Renal function markers | 48 weeks up to 96 weeks
  Serum creatinine, eGFR, uine beta-2 microglobulin, tubular resorption rate of phosphate, urine albumin, N-acetyl-beta-glucosaminidase, serum cystatin C, urine protein and urine glucose
Lipids | 48 weeks up to 96 weeks
  Triglycerides, HDL cholesterol, LDL cholesterol and total cholesterol
Adverse events | 96 weeks
  Adverse events of each arm, symptoms and rate
Blood plasma concentration of RAL and DRV | 96 weeks
  Blood plasma concentration level of raltegravir and darunavir among all consented and intervened cases at National Center for Global Health and Medicine
Discontinuation rate | 96 weeks
  Discontinuation rate of each arm, reason and timing

CONTACTS AND LOCATIONS:
Overall Officials: Shinichi Oka, MD PhD, Principal Investigator — National Center for Global Health and Medicine
Locations (1):
- National Center for Global Health and Medicine, Shinjuku, Tokyo, Japan

REFERENCES:
- [Result] Nishijima T, Gatanaga H, Shimbo T, Komatsu H, Endo T, Horiba M, Koga M, Naito T, Itoda I, Tei M, Fujii T, Takada K, Yamamoto M, Miyakawa T, Tanabe Y, Mitsuya H, Oka S; SPARE study team. Switching tenofovir/emtricitabine plus lopinavir/r to raltegravir plus Darunavir/r in patients with suppressed viral load did not result in improvement of renal function but could sustain viral suppression: a randomized multicenter trial. PLoS One. 2013 Aug 8;8(8):e73639. doi: 10.1371/journal.pone.0073639. eCollection 2013. PMID 23951362